CLINICAL TRIAL: NCT04963062
Title: Randomized Clinical Trial Evaluating the Efficiency and Safety of Holmium Laser With Moses Technology Versus SuperPulsed Laser System With Thulium Laser on Renal and Ureteral Stones
Brief Title: Moses vs. Thulium Laser Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-0695; A539800 (Other: UW Madison); SMPH/UROLOGY/UROLOGY (Other: UW Madison); Protocol ver 11-29-2021 (Other: HS-IRB UW Madison)
Record Dates: First submitted 2021-07-06; First posted 2021-07-15 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Urinary Tract Stone
Keywords: Lithotripsy; Holmium laser
MeSH Terms: conditions — Urinary Calculi | interventions — Lasers, Solid-State

STUDY DESIGN:
Intervention Model Description: Participants will be randomized (ratio 1:1) at the time of enrollment to be treated with either the holmium laser with Moses or the thulium laser. Investigators will use Permuted Block Randomization (stratified by stone size 3 - 10 mm or 11-20 mm) (block size 4).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Participants treated with Holmium laser with the Moses laser (Experimental)
  Interventions: Device: Holmium laser with Moses lasers
- Participants treated with Holmium laser with the thulium laser (Experimental)
  Interventions: Device: Holmium laser with thulium lasers

INTERVENTIONS:
Device: Holmium laser with Moses lasers — The holmium laser with Moses is FDA approved. It emits two separate laser pulses with a short time interval between them. The first pulse divides the water between the laser fiber tip and the stone and the second pulse hits the stone unobstructed. The goal is to increase stone ablative volume and decrease retropulsion of the stone.
  Arms: Participants treated with Holmium laser with the Moses laser
Device: Holmium laser with thulium lasers — The holmium laser with thulium laser is FDA approved. It has a different wavelength then the holmium laser with Moses and thus has slightly different energy properties. It has also been shown to increase ablative volume and decrease retropulsion without any safety concerns
  Arms: Participants treated with Holmium laser with the thulium laser

SUMMARY:
The incidence of urinary tract stone disease is increasing. According to the National Health and Nutrition Examination Survey, as of 2012, 10.6% of men and 7.1% of women in the United States are affected by renal stone disease. This has led to an increased demand on Urologists for efficient and safe surgical treatment of stone disease. Over the past two decades, ureteroscopy with laser lithotripsy has become the treatment of choice for most ureteral and renal stones globally. The holmium laser is considered the gold standard for laser lithotripsy. Holmium laser lithotripsy with Moses and the thulium laser are new technologies meant to improve the efficiency of laser lithotripsy. Both are FDA approved treatment modalities for stone disease. Two in vitro studies have compared Moses versus thulium and shown that thulium has higher ablative volumes then the holmium laser with Moses, but no clinical trials have compared the two treatment modalities.

In this study, investigators are going to conduct a prospective, randomized clinical trial to determine whether there is a difference in procedural time, intraoperative parameters or stone free rate between the Holmium laser with Moses and the thulium laser. This is significant as this may lead to shorter overall operative times, which may result in decreased operative costs and complications.

ELIGIBILITY:
Inclusion Criteria:

* Participants with renal or ureteral urinary stones who require endoscopic treatment in the outpatient operating room
* Participant's stone size in a single renal unit of 3-10 mm and 11-20 mm. Stone size is defined as the largest diameter of a single stone on pre-operative CT. Participants with multiple stones will be included as long as their largest stone size falls within the above parameters.

Exclusion Criteria:

* Participants under 18 years of age and over 89 years old.
* Pregnant participants
* Participants with transplant kidneys
* Participants with irreversible coagulopathy
* Participants with known ureteral stricture disease
* Participants who do not have a pre-operative CT.
* Non-English speaking, vulnerable participants such as lacking of decision-making capability, prisoner, adult unable to consent, will not be enrolled.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2023-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Nakada, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants Treated With Holmium Laser With the Moses Laser | Participants Treated With Holmium Laser With the Thulium Laser
Started | 56 | 58
Completed | 52 | 56
Not Completed | 4 | 2
Not completed — withdrew by the study team | 4 | 2

BASELINE CHARACTERISTICS:
Population: Patients withdrew were not included in the following data collection and analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants Treated With Holmium Laser With the Moses Laser | Participants Treated With Holmium Laser With the Thulium Laser | Total
Number analyzed (Participants) | 52 | 56 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 36 | 69
  >=65 years | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (12.8) | 59.6 (11.3) | 60.3 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 29 | 50
  Male | 31 | 27 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 50 | 56 | 106
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 52 | 55 | 107
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Procedural Time (Minutes)
Description: Time from the minute the ureteroscope is inserted into the participant to the time the ureteroscope has been removed will be reported as procedural time.
Time Frame: up to 6 hours
Measure: Median (Full Range); unit: minutes
Arm/Group | Participants Treated With Holmium Laser With the Moses Laser | Participants Treated With Holmium Laser With the Thulium Laser
Number analyzed (Participants) | 52 | 56
minutes | 20 [11 to 28] | 17 [13 to 24]

2. Secondary Outcome: Stone Free Rate
Description: Stone free rate (SFR) (%) are defined as either the absence of any residual stone fragments or the presence of clinically insignificant residual stone fragments in the urinary tract which were defined as ≦ 4mm, asymptomatic, non-obstructive and non-infectious stone particles.
Time Frame: Baseline(pre-operative) and approximately 8 weeks
Population: patients who did not have post operative image were not able to access stone free rate
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Treated With Holmium Laser With the Moses Laser | Participants Treated With Holmium Laser With the Thulium Laser
Number analyzed (Participants) | 47 | 53
Participants | 40 | 40

3. Secondary Outcome: Lasing Time (Minutes)
Description: Time the laser was in use, not including pedal pauses
Time Frame: up to 6 hours
Measure: Median (Full Range); unit: minutes
Arm/Group | Participants Treated With Holmium Laser With the Moses Laser | Participants Treated With Holmium Laser With the Thulium Laser
Number analyzed (Participants) | 52 | 56
minutes | 2.7 [1.2 to 6.7] | 3.6 [1.7 to 7.3]

4. Secondary Outcome: Total Energy Used (Kilojoules)
Description: The total energy used to fragment the stones into small pieces (≤2 mm)
Time Frame: up to 6 hours
Measure: Median (Full Range); unit: KJ
Arm/Group | Participants Treated With Holmium Laser With the Moses Laser | Participants Treated With Holmium Laser With the Thulium Laser
Number analyzed (Participants) | 52 | 56
KJ | 1.2 [0.5 to 4.7] | 2.5 [1.4 to 5.6]

5. Secondary Outcome: Ablation Efficiency (J/mm^3)
Description: It is a ratio of ablated stone volume to the laser pulse energy (J/mm3)
Time Frame: up to 6 hours
Measure: Median (Full Range); unit: J/mm^3
Arm/Group | Participants Treated With Holmium Laser With the Moses Laser | Participants Treated With Holmium Laser With the Thulium Laser
Number analyzed (Participants) | 52 | 56
J/mm^3 | 1.5 [0.7 to 2.2] | 1.8 [1.1 to 3.2]

6. Secondary Outcome: Number of Participants With Post-operative Complications
Time Frame: approximately 8 weeks (1 month post-operative)
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Treated With Holmium Laser With the Moses Laser | Participants Treated With Holmium Laser With the Thulium Laser
Number analyzed (Participants) | 52 | 56
Participants | 5 | 6

7. Secondary Outcome: Change in Quality of Life Survey (WISQOL Short Form) Both Pre-operatively and Post-operatively
Description: WISQOL short form is a 6 item questionnaire which can be scored from 1(worst outcome) to 5 (best outcome). The raw score range is 5-30. In the study, standardized total score is used. the range of the standardized total score is 0-100.
Time Frame: Baseline(pre-operative) and approximately 8 weeks (1 month post-operative)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Participants Treated With Holmium Laser With the Moses Laser Pre Operative Score: Quality of life assessment before treatment for patients treated with moses laser.
- Participants Treated With Holmium Laser With the Thulium Laser Pre Operative Score: Quality of life assessment before treatment for patients treated with thulium laser.
- Participants Treated With Holmium Laser With the Moses Laser Post Operative Score: Quality of life assessment after treatment for patients treated with moses laser.
- Participants Treated With Holmium Laser With the Thulium Laser Post Operative Score: Quality of life assessment after treatment for patients treated with thulium laser.
Arm/Group | Participants Treated With Holmium Laser With the Moses Laser Pre Operative Score | Participants Treated With Holmium Laser With the Thulium Laser Pre Operative Score | Participants Treated With Holmium Laser With the Moses Laser Post Operative Score | Participants Treated With Holmium Laser With the Thulium Laser Post Operative Score
Number analyzed (Participants) | 52 | 56 | 52 | 56
score on a scale | 51.5 (32.6) | 49 (33.1) | 75.3 (33.1) | 84.3 (19.1)

8. Secondary Outcome: Score on the Laser Evaluation Instrument
Description: Physician evaluation of the laser will be done by Laser Evaluation Instrument. It consists of 6 items which can be scored from 0(worst outcome) to 5 (best outcome). Cumulative score may range from 0-30.
Time Frame: Up to 6 hours
Population: Evaluation of the efficiency of the two lasers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants Treated With Holmium Laser With the Moses Laser | Participants Treated With Holmium Laser With the Thulium Laser
Number analyzed (Participants) | 52 | 56
score on a scale | 4.3 (0.5) | 4.5 (0.5)

9. Secondary Outcome: Ablation Speed
Description: The speed to fragment or dust stones
Time Frame: 0-6 hours
Measure: Median (Full Range); unit: mm^3 per minute
Arm/Group | Participants Treated With Holmium Laser With the Moses Laser | Participants Treated With Holmium Laser With the Thulium Laser
Number analyzed (Participants) | 52 | 56
mm^3 per minute | 482 [205 to 868] | 413 [273 to 692]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Participants Treated With Holmium Laser With the Moses Laser | Participants Treated With Holmium Laser With the Thulium Laser
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/56
Other Adverse Events (participants affected / at risk) | 5/52 | 6/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Treated With Holmium Laser With the Moses Laser (N=52) | Participants Treated With Holmium Laser With the Thulium Laser (N=56)
Obstructing fragments required surgical treatment (Renal and urinary disorders) | 1 (1) | 2 (2) — Patients had obstructing fragments which required unplanned surgery.
Obstructing fragments passed (Renal and urinary disorders) | 1 (1) | 0 (0) — Obstructing fragments passed successfully
ER visit and discharge (Renal and urinary disorders) | 1 (1) | 3 (3) — Patient ER visit within the follow up period
UTI treated with outpatient antibiotics (Renal and urinary disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT04963062/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT04963062/SAP_001.pdf